CLINICAL TRIAL: NCT02185053
Title: A Phase II, Single-Blind, Placebo-Controlled, Sequential Treatment, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of CPC-201 in Patients With Alzheimer's Disease Type Dementia
Brief Title: A Phase II Study of CPC-201 to Treat Alzheimer's Disease Type Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chase Pharmaceuticals Corporation, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPC-001-07
Record Dates: First submitted 2014-07-07; First posted 2014-07-09 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPC-201 (Experimental)
  Interventions: Drug: CPC-201

INTERVENTIONS:
Drug: CPC-201

SUMMARY:
This is a Phase II, Single-Blind, Placebo-Controlled, Sequential Treatment, Multiple Ascending Dose Study to Evaluate the Safety and Tolerability of CPC-201 in Patients with Alzheimer's Disease Type Dementia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 - 79 years inclusive.
* Meeting the diagnosis of probable Alzheimer's Disease
* Of moderate severity (Mini-Mental Status Exam [MMSE] score 10 - 20 inclusive).
* Patients must be in generally good health as indicated by their medical history and physical examination, vital signs, electrocardiogram (ECG), and standard laboratory tests.

Exclusion Criteria:

* Women of child bearing potential.
* History or presence of a seizure disorder.
* History of peptic ulcer disease, urinary or gastric retention; asthma or obstructive pulmonary disease.
* History or presence of bladder outflow obstruction, gastrointestinal obstructive disorder or reduced GI motility, or narrow-angle glaucoma.
* History or presence of gastrointestinal, hepatic, or renal disease, or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* History or presence of myasthenia.
* Known hypersensitivity to donepezil, solifenacin or related drugs.
* Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives.
* Patients who have participated in another clinical trial with an investigational drug within previous 30 days.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn James, Study Director — Allergan
Locations (1):
- CPC1, West Palm Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Solifenacin Dose Escalation: Solifenacin upward dose titration from 10 mg/day to 15 mg/day (together with donepezil 10 mg/day)
- Donepezil Dose Escalation: Donepezil upward dose titration up to the first intolerable dose (FID) or up to 40 mg/kg together with solifenacin 15 mg/day. End of dose escalation phase.
- Donepezil Dose Maintenance: Donepezil upward dose titration up to the first intolerable dose (FID) or up to 40 mg/kg together with solifenacin 15 mg/day. End of Dose Maintenance phase.
Period: Solifenacin Dose Escalation Phase
Arm/Group | Solifenacin Dose Escalation | Donepezil Dose Escalation | Donepezil Dose Maintenance
Started | 41 | 0 | 0
Completed | 38 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Cardiac symptoms | 1 | 0 | 0
Not completed — No longer meeting eligibility criteria | 2 | 0 | 0
Period: Donepezil Dose Escalation Phase
Arm/Group | Solifenacin Dose Escalation | Donepezil Dose Escalation | Donepezil Dose Maintenance
Started | 0 | 38 | 0
Completed | 0 | 33 | 0
Not Completed | 0 | 5 | 0
Not completed — Cardiac symptoms | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — No longer meeting eligibility criteria | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Donepezil Dose Maintenance Phase
Arm/Group | Solifenacin Dose Escalation | Donepezil Dose Escalation | Donepezil Dose Maintenance
Started | 0 | 0 | 33
Completed | 0 | 0 | 30
Not Completed | 0 | 0 | 3
Not completed — Cardiac symptoms | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All subjects who received at least one dose of any study drug.
Arm/Group | Safety Population
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Donepezil Maximum Tolerated Dose (MTD)
Description: Number of participants who reached Donepezil Maximum Tolerated Dose of 40 mg/day (highest allowed per protocol) at the end of donepezil dose titration phase and at the end of the maintenance phase.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Donepezil Dose Escalation | Donepezil Dose Maintenance
Number analyzed (Participants) | 33 | 33
Participants
  15 mg/day | 0 | 0
  20 mg/day | 0 | 0
  25 mg/day | 2 | 2
  30 mg/day | 1 | 2
  35 mg/day | 1 | 1
  40 mg/day | 29 | 28

2. Secondary Outcome: Number of Subjects With Any TEAEs
Description: Number of subjects who experienced any treatment-emergent adverse events (TEAEs) at any time during the study.
Time Frame: 6 months
Population: All subjects those who received at least one dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | Safety Population
Number analyzed (Participants) | 41
Participants
  Serious Adverse Events (SAEs) | 8
  Non-serious AEs | 34
  Deaths | 1

3. Secondary Outcome: Donepezil Plasma Concentration at Maximum Tolerated (MTD) or Maximum Allowable Dose
Description: Donepezil Plasma Concentration pre-dose and 4 hour post-dose at Maximum Tolerated (MTD) or Maximum Allowable Dose, measured at baseline, at end of donepezil dose titration and at the end of maintenance.
Time Frame: Day 1 (baseline) to end of study
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Solifenain Dose Escalation: Solifenacin upward dose titration from 10 mg/day to 15 mg/day (together with donepezil 10 mg/day)
Arm/Group | Solifenain Dose Escalation | Donepezil Dose Escalation | Donepezil Dose Maintenance
Number analyzed (Participants) | 41 | 32 | 29
ng/mL
  Donepezil Concentration pre-dose (ng/mL) | 42.7 (20.27) | 184.2 (65.95) | 188.1 (64.21)
  Donepezil Concentration 4 hour post-dose (ng/mL) | 57.2 (21.58) | 257.5 (80.56) | 269.2 (80.94)

ADVERSE EVENTS:
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 8/41
Other Adverse Events (participants affected / at risk) | 33/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=41)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Gastric volvulus (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=41)
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Fall (Injury, poisoning and procedural complications) | 5
Decreased appetite (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.